CLINICAL TRIAL: NCT06522841
Title: 16SRDNA Sequencing of 30 Samples of Human Oral Microbial Samples by Tianjin Medical University: Analysis of the Microbial Community Diversity in Various Regions of the Healthy Oral Cavity
Brief Title: 16SRDNA Sequencing of 30 Samples of Human Oral Microbial Samples by Tianjin Medical University
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Yuchang Liu, Department of Endodontics and Laboratory for Dental Stem Cells and Endocrine Immunology, Tianjin Medical University School of Stomatology, Tianjin, China., Tianjin Medical University
Other Study IDs: TMUhMEC20221105
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Oral Microbiome; Sampling Methods; Epidemiological Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Objective:

To explore suitable sampling sites and methods for oral epidemiological surveys in large populations, we aim to compare the distribution of the oral core microbiome at different sites and using different sampling methods in a small sample of healthy individuals.

Main Question:

What is the distribution of the oral core microbiome at different sampling sites and using different sampling methods in orally healthy individuals?

Study Design:

Participants will be randomly selected from a population of orally healthy individuals. After explaining the study to the participants and obtaining informed consent, they will complete a consent form and be informed of the precautions. Samples will be collected using cotton swabs and curettes from the buccal surface of the lower right first molar and using cotton swabs from the left and right buccal mucosa. The samples will be placed in pre-numbered test tubes and sent to the laboratory for microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

* (1) People who had no oral diseases particularly caries, periodontitis, and oral mucosal diseases. (2) Teeth without previous restorations.

Exclusion Criteria:

* (1) People who are pregnant. (2) People who suffer from severe systematic diseases, such as diabetes, immune system diseases, and genetic diseases. (3) People who have taken antibiotics within two weeks before sampling.(4) People who have had or currently receiving radiotherapy or chemotherapy. (5) People with complete or incomplete absence of dentition. (6) Individuals who smoke or have smoked within the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to WHO-related standards, we have selected adults who are orally healthy, free from systemic diseases, and non-smokers.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
16SRDNA sequencing of 30 samples of human oral microbial samples by Tianjin Medical University | 2021.07 - 2021.12 Finalize research topic. 2021.12 - 2022.06 Complete bibliometric analysis. 2022.06 - 2022.12 Acquire data for analysis. 2022.12 - 2023.06 Obtain analysis results. 2023.06 - 2024.01 Complete and submit the thesis.
  Four sites were assessed: the buccal mucosa on both sides and the buccal surfaces of the left and right mandibular first molars. Two sampling methods, swab and curette, were used to collect bacterial communities from healthy individuals. Specifically, buccal mucosa samples (n=10) and tooth surface samples (n=20) were analyzed using 16S rDNA gene sequencing. Bacterial signals were detected through fluorescence in situ hybridization (FISH), targeting the bacterial 16S rDNA gene. Metastats analysis and Wilcoxon test were used.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University School of Stomatology, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Objective:
  Our goal is to facilitate the advancement of scientific research by sharing individual participant data (IPD) from our study on the microbial community diversity in various regions of the healthy oral cavity. This sharing plan is designed to ensure that data is accessible to researchers while protecting the privacy and confidentiality of study participants.
  Data to be Shared:
  The IPD to be shared includes:
  1. Demographic Information:
     * Age
     * Gender
  2. Microbial Data:
     * Microbiome sequencing data (raw and processed sequences)
     * Operational Taxonomic Units (OTUs) and species-level identification
  3. Sampling and Processing Details:
     * Method of sample collection (swab vs. scraper)